CLINICAL TRIAL: NCT04491578
Title: Effects of an Advance Care Planning Programme for Persons With Early Stage Dementia in the Community: A Quasi-experimental Study
Brief Title: An Advance Care Planning Programme for Persons With Early Stage Dementia in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Collaborators: Chinese University of Hong Kong (Other); Food and Health Bureau, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Ms Cheryl Yeung Chi Yan, Senior Lecturer, Hong Kong Metropolitan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HMRF 03180198
Record Dates: First submitted 2020-06-06; First posted 2020-07-29 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Dementia Mild; Mild Cognitive Impairment
Keywords: advance care planning
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Dyads of participants recruited from all elderly community centres will receive the ACP intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACP programme (Experimental): It is a theory-driven ACP programme specifically designed for PWEDs or persons with MCI and their family caregivers. The intervention is underpinned by the Bandura's self-efficacy model and shared decision-making model.
  Interventions: Behavioral: ACP programme "Have a Say"

INTERVENTIONS:
Behavioral: ACP programme "Have a Say" — Each dyad of participants will receive a 4-session ACP programme, which consists of educational components, guided reflection, and dyadic ACP discussion, guided by ACP facilitators and an ACP booklet. It is composed of 2 group-based sessions and 2 dyadic discussions. One hour for each session. The group-based sessions are nurse-led, in which dyads of participants will be provided with information about the trajectory of dementia, their future healthcare needs and caring options. Their values and care preferences on future care will be elicited in a consistent manner. The dyadic sessions are led by trained ACP facilitator. Dyads of participants will be supported to have an individualized ACP discussion. By the end of the programme, each dyad of participants will be given an ACP booklet documenting the ACP process.

SUMMARY:
Advance care planning (ACP) has been widely advocated for persons with early stage dementia (PWEDs) and persons with mild cognitive impairment (MCI). This proposed study attempts to promote the uptake of ACP for this population and their family caregivers in the community and to examine the effects of an ACP programme "Have a Say" for this population. It is hypothesized that participants received the intervention will be more engaged in ACP and their dyadic concordance on end-of-life care preference with their family caregivers will be higher after the intervention.

DETAILED DESCRIPTION:
This study aims to evaluate the impacts of an advance care planning (ACP) programme "Have a Say" for persons with early stage dementia (PWEDs) or MCI and their family caregivers in the community. A quasi-experimental study with repeated blinded outcome assessment will be conducted to assess the effects of an ACP programme on dyads of PWEDs or persons with MCI and their family caregivers recruited from elderly community centres. Individuals who have a clinical diagnosis of any form of dementia at the early stage or MCI or have a Global Deterioration Score (GDS) 3 or 4 will be eligible to this study. Participants will receive a 4-session ACP programme. It includes an educational component, guided reflection and ACP discussion through a series of group-based activity and dyadic discussion delivered by trained ACP facilitator and guided by an ACP booklet. Dyads of participants will be provided with information about the trajectory of dementia, their future healthcare needs and caring options. Their values and care preferences on future care will be elicited in a consistent manner. They will be supported to have an individualized ACP discussion. The primary study outcome is the ACP engagement level of PWEDs. Secondary outcome is the dyadic concordance on end-of-life care preference. Adverse outcomes such as depression and caregivers' burden will also be evaluated. Data collection will be conducted at baseline, immediately after, and one-month after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* aged 55 years or over;
* being Chinese,
* being a Cantonese speaker,
* having a Global Deterioration Scale score 3 or 4,
* having a designated family caregiver willing to participate in this study

Exclusion Criteria:

* non-communicable,
* mentally incompetent,
* received an ACP intervention,
* have previously signed an advance directive,
* have other life-limiting chronic illnesses with a life expectancy of less than 6 months.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-01-09 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Change in advance care planning engagement | Baseline, immediately after the intervention, 1 month follow up
  The behavior change process in ACP behaviours is measured using a 9-item ACP engagement survey. It covers two sub-scales, self-efficacy and readiness, of ACP engagement. Each item is rated on a 5-point likert scale. The higher score means the higher level of engagement for the ACP behaviour.

SECONDARY OUTCOMES:
Change in dyadic concordance of end-of-life care preferences | Baseline, immediately after the intervention, 1 month follow up
  The dyadic concordance on end-of-life care preferences is measured by a modified Life Support Preferences Questionnaire (LSPQ). Dyads of participants are invited to answer individually, simultaneously but separately for a hypothetical scenario featured the prospect of developing into advanced stage of dementia. PWEDs are asked to indicate their preference for receiving three discrete life-sustaining medical treatments (cardio-pulmonary resuscitation, mechanical ventilation and tube feeding) using a 3 point Likert Scale (1=want to attempt; 2=refuse; 3= not sure). The dyadic congruence is determined based on whether both of them choose the same option for end-of-life treatments, regardless that was for active treatment or not, they gained a score of one. Given the nature of ACP is for the dyad to communicate preferences on end-of-life care, no score would be given if anyone in the dyad chose the "not sure" response.

OTHER OUTCOMES:
Depression | Baseline, immediately after the intervention, 1 month follow up
  The level of depression of PWEDs is measured by the 19-item Cornell Scale for Depression in Dementia (CSDD). It is to evaluate any adverse outcome posed by the intervention on them.
Caregivers' stress | Baseline, immediately after the intervention, 1 month follow up
  Caregivers' stress is measured by the 12-item Zarit Caregiver Burden Interview. It is to evaluate any adverse outcome posed by the intervention on family caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Yan Cheryl Yeung, MN, Principal Investigator — Chinese University of Hong Kong
Locations (10):
- Hong Kong (10):
  - HKSKH Lok Man Alice Kwok Integrated Service Centre, Kowloon
  - Hong Kong Christian Service, Kowloon
  - Yang Memorial Methodist Social Service Choi Hung Community Centre for Senior Citizens, Kowloon
  - The Neighbourhood Advice-Action Council Sham Shui Po District Elderly Community Centre, Sham Shui Po
  - Jockey Club Centre for Positive Ageing, Shatin
  - The Neighbourhood Advice- Action Council Ma On Shan Neighbourhood Elderly Centre, Shatin
  - The Neighbourhood Advice-Action Council Tuen Mun District Integrated Services Centre for the Elderly, Tuenmen
  - Yau On Lutheran Centre for the Elderly, Tuenmen
  - HKSKH Chuk Yuen Canon Martin District Elderly Community Centre, Wong Tai Sin
  - Pentecostal Church of Hong Kong Ltd.Choi Wan Neighbourhood Elderly Centre, Wong Tai Sin

IPD SHARING:
Plan to Share IPD: No